CLINICAL TRIAL: NCT00962988
Title: Efficacy and Cost-effectiveness of Cost-free Pharmacotherapy for Smoking Cessation for High-risk Smokers With Cerebrovascular Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIPRC-6749
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Cerebrovascular Disorders; Smoking Cessation
Keywords: Cerebrovascular disease; stroke; Transient Ischemic Attack; smoking cessation; Pharmacotherapy
MeSH Terms: conditions — Cerebrovascular Disorders; Smoking Cessation; Stroke; Ischemic Attack, Transient | interventions — Tobacco Use Cessation Devices; Varenicline; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cost-Free Group (Experimental)
  Interventions: Drug: Cost-Free Pharmacotherapy Group
- Prescription Only Group (Other)
  Interventions: Other: Prescription Only Group

INTERVENTIONS:
Drug: Cost-Free Pharmacotherapy Group — Participants assigned to the cost-free pharmacotherapy group will be provided with a 12-week supply of NRT, or a 12-week supply of bupropion or varenicline.
  Patients smoking 10 cigarettes or less will be prescribed 7mg/24hours for 12 weeks. Those who smoke 11- 20 cigarettes per day will be prescribed 14 mg/24 hours for 8 weeks and then nicotine patch 7mg for 4 weeks. Those smoking ≥ 20 cigarettes per day will be prescribed 21 mg/daily for 6 weeks and then nicotine patch 14mg/daily for 4 weeks and then nicotine patch 7 mg/daily for 2 weeks.
  For patients who are prescribed varenicline, they will start the medication 8 days before the quit date using the following regime: Days 1-3: 0.5mg once/day; Days 4-7: 0.5 mg BID; Day 8-12 weeks 1.0 mg twice daily.
  For patients who are prescribed bupropion, they will start the medication 8 days before the quit date using the following regime: Days 1-3: 150 mg daily (in the morning); Day 4-30: 150 mg BID for 3 months.
  Other Names: Nicotine Patch; Champix; Chantix; Wellbutrin
  Arms: Cost-Free Group
Other: Prescription Only Group — Participants assigned to the prescription only usual care group will be asked to have their prescription for smoking cessation pharmacotherapy filled at their own cost at their local community pharmacy
  Arms: Prescription Only Group

SUMMARY:
Research Aims

The aims of this research study are to determine whether cost-free smoking cessation pharmacotherapy:

1. Helps smokers with Transient Ischemic Attack (TIA) or stroke to quit smoking over the long-term, compared to simply providing a prescription for these medications;
2. Is a more cost-effective alternative to providing a prescription only for these medications in this high risk population.

Hypotheses to be Tested

The hypotheses to be tested include the following:

1. The CO-validated continuous abstinence rate at weeks 26 and 52 following a target quit date will be at least 10% higher for the cost-free smoking cessation pharmacotherapy intervention group compared to the prescription only usual care group;
2. Cost-free smoking cessation pharmacotherapy will have a greater cost-effectiveness (i.e., cost/quit) than providing a prescription only.

DETAILED DESCRIPTION:
Smokers with Transient Ischemic Attack (TIA) or stroke attending a Stroke Prevention Clinic and willing to quit smoking will be randomly assigned (1:1) to either a prescription only (PO) usual care group or a cost-free (CF) pharmacotherapy experimental group. Participants assigned to the prescription only usual care group will be asked to have their prescription for smoking cessation pharmacotherapy filled at their own cost at their local community pharmacy. Participants assigned to the cost-free pharmacotherapy group will be provided with a 12-week supply of NRT, or a 12-week supply of bupropion or varenicline. The pharmacotherapy will be provided by the research nurse to the patient immediately. All participants will receive identical advice regarding smoking from the attending neurologist, nurse counseling for smoking cessation, and follow-up tracking and telephone-based support for up to 26 weeks after the target quit date. Non-treatment follow-up will continue to week 52 after the target quit date.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a current daily smoker (one cigarette per day in the month preceding the visit to the Stroke Prevention Clinic)
2. Patient has been diagnosed with TIA or stroke at any point in time
3. Patient is able, in the opinion of the neurologist, to comprehend and participate in the smoking cessation interventions
4. Patient is 18 years of age or older
5. Patient is willing to set a quit date
6. Patient willing to travel to study centre for follow-up visits
7. Patient is willing to provide informed consent

Exclusion Criteria:

1. Patient is unable to understand English or French
2. Patient is not willing to use pharmacotherapy to quit
3. Patient has been using smoking cessation medication for more than 6 weeks directly prior to clinic visit or hospital admission.
4. Patient is pregnant, lactating or planning to become pregnant during the study period
5. Patient has contraindication(s) to all of the following smoking cessation medications:

   * Nicotine replacement therapy (allergy to adhesive, serious cardiac arrhythmias (e.g., tachycardia), vasospastic disease (e.g., Buerger's disease, Prinzmetal's variant angina)
   * Bupropion (history of seizure disorder or head trauma; presently taking Wellbutrin; previous reaction to bupropion/Zyban/Wellbutrin; pre-existing or current eating disorder; taking anti-depressants, antipsychotics, corticosteroids, MAO inhibitors, theophylline, cocaine or diet pills; taking a quinalone antibiotic (e.g., ciprofloxacin, levoflozacin); currently using oral hypoglycemic product or insulin; severe hepatic impairment; CNS tumour; and
   * Varenicline (renal failure; use of cimetidine; previous reaction to varenicline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2009-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the biochemically confirmed (exhaled CO < 10 ppm) self-reported continuous abstinence from weeks 12 to 52 following the target quit date. | 52 weeks

SECONDARY OUTCOMES:
The secondary outcome will be the biochemically confirmed (exhaled CO < 10 ppm) self-reported continuous abstinence from weeks 12 to 26 following the target quit date. | 26 weeks
The total costs of smoking cessation treatment will be tracked over the duration of the study to determine the cost-effectiveness of providing cost-free pharmacotherapy for smoking cessation versus a prescription only. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Grant Stotts, MD, Principal Investigator — The Ottawa Hospital; Andrew Pipe, MD, Study Chair — Ottawa Heart Institute Research Corporation; Sophia Papadakis, MHA, Study Chair — Ottawa Heart Institute Research Corporation; Debbie Aitken, RN BScN, Study Chair — Ottawa Heart Institute Research Corporation; Kerri-Anne Mullen, MSc, Study Chair — Ottawa Heart Institute Research Corporation; Sophia Gocan, RN BScN, Study Chair — The Ottawa Hospital; Mary Ann Laplante, RN BScN, Study Chair — The Ottawa Hospital; Robert Reid, MBA PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (2):
- Canada (2):
  - Hamilton Health Sciences -Stroke Prevention Clinic, Hamilton, Ontario
  - The Ottawa Hospital - Stroke Prevention Clinic, Ottawa, Ontario